CLINICAL TRIAL: NCT04205526
Title: Canadian Platform for Trials With Non-Invasive Brain Stimulation: Contralesional Inhibitory rTMS for Recovery of Arm Function After Stroke - A Feasibility Trial (Canstim: ConTRA-Stroke-F)
Brief Title: Contralesional Inhibitory rTMS for Recovery of Arm Function After Stroke
Acronym: ConTRAstroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thiel, Alexander, M.D. (Individual)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Dr. Alexander Thiel, Neurologist, Researcher, Thiel, Alexander, M.D.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MP-05-2020-1891
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Feasibility Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The only individual that will be unblinded is the person administering the rTMS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Experimental): Sub-acute stroke patients will be randomized to receive actual rTMS treatment. 1Hz rTMS will be applied over contralesional M1 at an intensity of 120% resting motor threshold once daily for 30 minutes (approximately 1800 pulses) for a total of 15 sessions.
  Interventions: Device: Active rTMS
- Sham control (Sham Comparator): Sub-acute stroke patients randomized to receive sham rTMS. For sham-stimulation, the TMS coil will be placed over the inter-hemispheric fissure at the vertex and stimulation will be performed with low intensity (10% resting motor threshold). This will cause similar skin sensations as real stimulation but will not induce currents in motor relevant areas.
  Interventions: Device: Sham TMS

INTERVENTIONS:
Device: Active rTMS — Patients randomized to receive actual rTMS treatment will receive 1Hz rTMS applied over contralesional M1 at an intensity of 120% resting motor threshold once daily for 30 minutes (approximately 1800 pulses) for a total of 15 sessions.
  Arms: Active rTMS
Device: Sham TMS — For sham-stimulation, the TMS coil will be placed over the inter-hemispheric fissure at the vertex and stimulation will be performed with low intensity (10% resting motor threshold). This will cause similar skin sensations as real stimulation but will not induce currents in motor relevant areas.
  Arms: Sham control

SUMMARY:
The CanStim consensus working group (multidisciplinary team of experts in rTMS from institutions across Canada) developed consensus recommendations for a protocol to deliver rTMS as an adjunct to physiotherapy to improve arm function in a Pan-Canadian stroke rehabilitation clinical trial. The overall goal of this multi-center feasibility trial is not to demonstrate that rTMS is effective, but to demonstrate that each site can recruit the assigned number of patients within a certain period, perform the stimulation procedure in conjunction with the protocol-specified physiotherapy intervention, complete the therapy protocol and enter complete datasets for each patient into the CanStim database. A secondary aim is to identify potential weaknesses of the consensus protocol that may need to be modified before performing a larger scale trial testing for the efficacy of the intervention.

DETAILED DESCRIPTION:
Rehabilitation is critical for reducing stroke-related disability. Although intensive physiotherapy improves function after a stroke, the frequency and intensity of therapy in a standard clinical rehabilitation session is insufficient to invoke these changes. Transcranial magnetic stimulation (TMS) is a safe, non-invasive method of stimulating the human brain. Repetitive TMS (rTMS) may have the potential to enhance the brain's ability to re-learn specific functions and reduce the amount of standard therapy required to achieve certain functional gains after stroke. Although two recent multicenter studies have begun to test the benefits of applying rTMS during stroke rehabilitation, large scale clinical trials demonstrating the efficacy of rTMS for post-stroke functional motor recovery are lacking. The use of rTMS interventions in stroke rehabilitation trials has been limited by a lack of consensus regarding the optimal protocol for the clinical application of TMS in stroke populations. The Canadian Platform for Trials in Non-Invasive Brain Stimulation (CanStim) is a national platform that aims to facilitate multicenter clinical trials for non-invasive brain stimulation interventions to augment recovery from stroke. As a first step, CanStim investigators convened a multidisciplinary team of experts in rTMS from institutions across Canada to form the CanStim Consensus Working Group and develop consensus recommendations for a protocol to deliver rTMS as an adjunct to standard therapy in a national stroke rehabilitation clinical trial.

ELIGIBILITY:
Inclusion Criteria: Stroke patients between 2 weeks and 3 months of stroke onset, patients with both cortical and subcortical stroke, age between 18 and 90 years, English or French as language of daily use, patients must be able to participate in a standard of care upper extremity therapy program and must be able to perform the GRASP AND should have a minimum deficit that they can improve (e.g., <= 56 on FM UE).

Exclusion Criteria: Prior symptomatic ischemic or hemorrhagic stroke, severe comprehension deficit that may compromise informed consent or understanding of instructions, contraindications to MRI and/or TMS, neurodegenerative or psychiatric disease, epilepsy or EEG-documented epileptic discharges, chronic renal or liver failure, life-threatening diseases limiting life expectancy to less than 6 months and auditory or visual deficits that cannot be corrected and might impair testing.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Fugl-Meyer Upper Arm Assessment between baseline, Post Day 1 and Post Day 30 | Baseline Testing done within the first three days then at 1 and 30 days post treatment. The Fugl Meyer has a minimum score of 0 and maximum score of 66. The higher the score the better the outcome.
  Index to assess sensorimotor impairment in stroke.
Change in the Action Research Arm Test between baseline, Post Day 1 and Post Day 30 | Baseline Testing done within the first three days then at 1 and 30 days post treatment. The test is scored from 0-57. The higher the score the better the outcome.
  An evaluative measure to assess specific changes in limb function among individuals who sustained cortical damage resulting in hemiplegia. It can assess a patients ability to handle objects differing in size, weight and shape and therefore can be considered to be an arm-specific measure of activity limitation.
Change in the Modified Rankin Scale between baseline, Post Day 1 and Post Day 30 | Baseline Testing done within the first three days then at 1 and 30 days post treatment. The scale is between 0-6. Zero being no symptoms to 6 the patient is dead. The lower the score the better the outcome.
  It is a scale for measuring the degree of disability or dependence in the activites of daily living in individuals who have suffered a stroke.

SECONDARY OUTCOMES:
Change in the Canadian Occupational Performance Measure between baseline, Post Day 1 and Post Day 30 | Baseline Testing done within the first three days then at 1 and 30 days post treatment. Two scores are obtained from each participant, one for performance and one for satisfaction. Each are scored between 0-10. The higher the value the better.
  This measure serves to identify issues of personal importance to the client and to detect changes in a client's self-perception of occupational performance over time.

CONTACTS AND LOCATIONS:
Overall Officials: ALEXANDER THIEL, MD, Phd, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No